CLINICAL TRIAL: NCT01705405
Title: Merging of Endoscopic and Ultrasound Images for Laparoscopic Surgery
Acronym: FEE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to a problem of device
Sponsor: AdministrateurCIC (Other)
Collaborators: TIMC-IMAG (Other); Clinical Investigation Centre for Innovative Technology Network (Network)
Responsible Party: Sponsor-Investigator, AdministrateurCIC, principal investigator, University Hospital, Grenoble
Organization: University Hospital, Grenoble (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: DCIC 12 06
Record Dates: First submitted 2012-10-05; First posted 2012-10-12 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Prostate Cancer
Keywords: cancer; prostate
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- medical device (Experimental): medical device to acquire ultrasound and endoscopic images during surgery
  Interventions: Device: Software for acquiring ultrasound and endoscopic images

INTERVENTIONS:
Device: Software for acquiring ultrasound and endoscopic images — Use of a medical device to acquire ultrasound and endoscopic images

SUMMARY:
Visualize surgical needles inserted in the prostate, under the ultrasound modality.

DETAILED DESCRIPTION:
In order to help the surgeon to remove the prostate during a laparoscopic intervention, our goal is to provide an innovative medical device that merges intra-operative ultrasound and endoscopic images.

We have already achieved the proof of concept of a device that merges ultrasound and endoscopic images. The objectives of this clinical trial are to accompany the maturation of the fusion device and to make the initial assessments of its Medical Service.

The main difficulty is to visualize markers (surgical needles) under both modalities , in order to merge them.

ELIGIBILITY:
Inclusion Criteria:

* of-age patient
* patient for whom a radical prostatectomy is planned
* patient with a prostate volume between 30g and 100g
* patient affiliated to the social security or equivalent
* Written informed consent

Exclusion Criteria:

* contraindication
* patient who has undergone a significant prostate resection
* patient who has undergone a prostate irradiation
* patient concerned by the L1121-6 à 8 of the health public code

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-10; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Percent of surgical needles visible under the ultrasound modality (once inserted in the prostate) | 1year

SECONDARY OUTCOMES:
Percent of data(ultrasound and endoscopic) on which the merging works | 1year
Percent of accurate merging | 1year
  the merging is accurate if its error is under 5mm
Percent of mistaken segmentation of the vesical neck in the endoscopic image | 1year
  The segmentation in the endoscopic image is mistaken if it differs of more than 5mm² from the segmentation in the ultrasound volume

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Alexandre Long, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Urology, University hospital of Grenoble, Grenoble, Isère, France

REFERENCES:
- See also: Related Info — http://www.cic-it-grenoble.fr/